CLINICAL TRIAL: NCT01975519
Title: A Phase 1B Dose-escalation and Phase 2a Study of Carotuximab (TRC105) in Combination With Pazopanib in Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105SAR101
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Advanced Soft Tissue Sarcoma
Keywords: TRC105; CD105; Endoglin; Angiogenesis Inhibitor; STS; Soft Tissue Sarcoma; TKI; Tyrosine Kinase Inhibitor; Pazopanib; Votrient; Advanced Soft Tissue Sarcoma; Angiosarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma | interventions — carotuximab; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRC105 and Pazopanib (Experimental): Weekly TRC105 in combination with standard dose pazopanib or every two week administration during cycle 1, and starting on cycle 2 day 1 and beyond, TRC105 may be administered every two weeks. This is also in combination with standard dose pazopanib.
  Interventions: Drug: TRC105 and Pazopanib

INTERVENTIONS:
Drug: TRC105 and Pazopanib — Weekly TRC105 in combination with standard dose Pazopanib.
  Other Names: Chimeric Antibody (TRC105) to CD105; Votrient

SUMMARY:
The purpose of the phase 1b portion is to evaluate safety and tolerability and determine a recommended phase 2 dose for TRC105 when added to standard dose pazopanib in patients with advanced soft tissue sarcoma. Up to 30 patients will be treated.

The purpose of the phase 2 portion is to estimate the PFS of patients with advanced soft tissue sarcoma by RECIST 1.1 and estimate ORR in a separate cohort of patients with angiosarcoma by RECIST 1.1. Up to 89 patients will be treated in phase 2, including two cohorts of up to 13 patients with angiosarcoma.

DETAILED DESCRIPTION:
Pazopanib is an oral inhibitor of multiple receptor tyrosine kinases, including vascular endothelial growth factor receptor VEGFR-1, VEGFR-2, and VEGFR-3 at therapeutic plasma concentrations. These receptors are implicated in pathologic angiogenesis, tumor growth, and cancer progression. Pazopanib is approved for the treatment of advanced soft tissue sarcoma, following progression on one prior systemic therapy, based on improved progression free survival. TRC105 is an antibody to CD105, an important angiogenic target on vascular endothelial cells that is distinct from VEGFR. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models and complements the activity of bevacizumab and multi-kinase inhibitors that target the VEGFR. In a phase 1 study of advanced solid tumors, TRC105 therapy caused a global reduction in angiogenic biomarkers and reduced tumor burden at doses that were well-tolerated. In a phase 1b study, the combination of TRC105 and bevacizumab produced radiographic reductions in tumor volume in bevacizumab-refractory patients, and was well tolerated. TRC105 potentiates bevacizumab and VEGFR tyrosine kinases (VEGFR TKI) in preclinical models. By targeting a non-VEGF pathway that is upregulated following VEGF inhibition, TRC105 has the potential to complement VEGFR TKIs and could represent a major advance in cancer therapy. Together, the use of TRC105 with pazopanib may result in more effective angiogenesis inhibition and improved clinical efficacy over that seen with pazopanib alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed unresectable soft tissue sarcoma that has progressed following treatment with chemotherapy. Prior pazopanib is allowed if the drug was not discontinued for toxicity ( Phase 1b only)
2. Histologically confirmed metastatic soft tissue sarcoma that has progressed by RECIST following treatment with anthracycline chemotherapy. Patients may have received up to four lines of systemic therapy for metastatic disease and no more than two lines of combination treatment ( Phase 2 only)
3. Histologically confirmed locally advanced (e.g. unresectable) or metastatic angiosarcoma that has progressed following treatment with prior systemic therapy. Progression must be documented on or following the most recent systemic therapy. Prior pazopanib is allowed if the drug was not discontinued for toxicity (Phase 2 angiosarcoma cohorts only)
4. Measurable disease by RECIST
5. Age of 12 years or older (patient must weigh ≥ 40 kg)
6. ECOG performance status ≤ 1
7. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade ≤ 1 or baseline (except alopecia or neuropathy)
8. Adequate organ function.
9. Willingness and ability to consent for self to participate in study
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
11. Available archival tumor specimen of the soft tissue sarcoma that meets inclusion criterion #1, #2 or #3

Exclusion Criteria:

1. Prior treatment with TRC105
2. Prior treatment with a VEGFR TKI (including pazopanib) (Phase 2 only)
3. Current treatment on another therapeutic clinical trial
4. Receipt of systemic anticancer therapy, including investigational agents, within 28 days of starting study treatment.
5. No major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure; date of surgery (if applicable) or the anticipated need for a major surgical procedure within the next six months.
6. Patients who have received wide field radiotherapy ≤ 28 days or limited field radiation for palliation < 14 days prior to cycle 1 day 1 or those patients who have not recovered adequately from side effects of such therapy
7. Uncontrolled chronic hypertension
8. Significant ascites or pericardial or pleural effusion
9. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
10. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, PTCA or CABG within the past 6 months. Deep venous thrombosis within 6 months, unless the patient is anti-coagulated without the use of warfarin for at least 2 weeks. In this situation, low molecular weight heparin is preferred.
11. Active bleeding or pathologic condition that carries a high risk of bleeding. Patients who have been uneventfully anti-coagulated with low molecular weight heparin are eligible.
12. Thrombolytic use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
13. Known active viral or nonviral hepatitis or cirrhosis
14. History of hemorrhage or hemoptysis within 3 months of starting study treatment
15. History of peptic ulcer within the past 3 months of treatment
16. History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved
17. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
18. Receipt of a strong CYP3A4 inducer within 12 days prior to cycle 1 day 1 or a strong CYP3A4 inhibitor within 7 days prior to cycle 1 day 1.
19. Pregnancy or breastfeeding. Female patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to first dose. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate.
20. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, Study Director — Tracon Pharmaceuticals Inc.
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sarcoma Oncology Center, Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai School of Medicine-Tisch Cancer Institute, New York, New York
  - Duke University, Durham, North Carolina
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- 8 mg/kg TRC105 + Pazopanib: 8 mg/kg of TRC105 in combination with standard dose pazopanib in patients with advanced soft tissue sarcoma.
- 10 mg/kg TRC105 + Pazopanib: 10 mg/kg of TRC105 in combination with standard dose pazopanib in patients with advanced soft tissue sarcoma.
Period: Overall Study
Arm/Group | 8 mg/kg TRC105 + Pazopanib | 10 mg/kg TRC105 + Pazopanib
Started | 3 | 108
Phase 1b | 3 | 23
Phase 2a Soft Tissue Sarcoma | 0 | 63
Phase 2a Angiosarcoma Cohort | 0 | 22
Completed | 3 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 mg/kg TRC105 + Pazopanib | 10 mg/kg TRC105 + Pazopanib | Total
Number analyzed (Participants) | 3 | 108 | 111
Age, Continuous [Median (Full Range); unit: years] | 55 [25 to 69] | 58 [19 to 89] | 58 [19 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 59 | 60
  Male | 2 | 49 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 6 | 6
  Black or African American | 1 | 8 | 9
  Caucasian | 2 | 89 | 91
  Hispanic or Latino | 0 | 5 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 108 | 111
ECOG Performance Status [Count of Participants; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all self care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. = Capable of only limited self care; confined to bed or chair more than 50% of waking hours
  4. = Completely disabled; cannot carry on any self care; totally confined to bed or chair
  5. = Dead
  Participants
    ECOG Grade 0 | 2 | 31 | 33
    ECOG Grade 1 | 1 | 77 | 78
    ECOG Grade 2 | 0 | 0 | 0
    ECOG Grade 3 | 0 | 0 | 0
    ECOG Grade 4 | 0 | 0 | 0
    ECOG Grade 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: For DLT evaluation, severity (grade) was classified according to common terminology criteria for adverse events version 4.0 (CTCAE v4.0). DLTs were defined as grade 4 neutropenia persisting for ≥ 5 days, febrile neutropenia (grade 4 neutropenia with fever > 38.5 ºC both sustained over a 24 hour period), neutropenic infection (grade ≥ 3 neutropenia with grade ≥ 3 infection), anemia ≥ grade 4, grade > 4 thrombocytopenia or grade ≥ 3 thrombocytopenia and grade ≥ 3 hemorrhage, or grade 3 or 4 nonhematologic toxicity with the following exceptions: nausea, vomiting, or diarrhea for <48 hours, asymptomatic electrolyte abnormalities that are corrected to grade 1 or better in < 72 hours, or headache lasting less than 48 hours.
Time Frame: 56 days
Population: All phase 1b patients who received at least a portion of a dose of TRC105
Measure: Count of Participants; unit: Participants
Groups:
- TRC105 Plus Pazopanib: All patients in Phase 1b portion of study who received TRC105 + Pazopanib TRC105: IV (8 mg/kg or 10 mg/kg). Pazopanib: oral (800 mg)
Arm/Group | TRC105 Plus Pazopanib
Number analyzed (Participants) | 26
Participants
  Patients with DLT at 8 mg/kg | 0
  Patients without DLT at 8 mg/kg | 3
  Patients with DLT at 10 mg/kg | 1
  Patients without DLT at 10 mg/kg | 22

2. Primary Outcome: Progression Free Survival of Patients With Advanced Soft Tissue Sarcoma (Phase 1 and 2)
Description: Number of patients with progression free survival, as defined as time from screening to either first disease progression or death from any cause per RECIST version 1.1
Time Frame: from screening to either disease progression or death
Population: All patients with scans completed at baseline and at least 1 time point on study.
Measure: Mean (95% Confidence Interval); unit: months
Groups:
- 8 mg/kg TRC105 + Pazopanib: All patients who received 8 mg/kg TRC105 + Pazopanib
- 10 mg/kg TRC105 + Pazopanib: All patients who received 10 mg/kg TRC105 + Pazopanib
Arm/Group | 8 mg/kg TRC105 + Pazopanib | 10 mg/kg TRC105 + Pazopanib
Number analyzed (Participants) | 3 | 90
months | 5.06 [4.96 to NA] — Not enough events to estimate an upper confidence level | 3.45 [2.56 to 3.85]

3. Primary Outcome: Objective Response Rate in a Cohort of Patients With Angiosarcoma
Description: The best response according to RECIST 1.1 for each patient in the phase 2 angiosarcoma cohort with measurable disease and who received at least one dose of study drug will be listed by cohort and tumor type
Time Frame: 1.5 years
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg/kg TRC105 + Pazopanib With Angiosarcoma: 10 mg/kg of TRC105 in combination with standard dose pazopanib in patients with advanced soft tissue sarcoma.
Arm/Group | 10 mg/kg TRC105 + Pazopanib With Angiosarcoma
Number analyzed (Participants) | 5
Participants
  Complete Response (CR) | 2
  Partial Response (PR) | 0
  Stable Disease (SD) | 3
  Progressive Disease (PD) | 0
  Not Evaluable | 0

4. Secondary Outcome: Trough Concentrations of TRC105 (Phase 2)
Description: Trough serum TRC105 concentrations will be measured using validated ELISA methods.
Time Frame: 4, 6, 8, and 10 weeks
Population: All patients who received at least a portion of a dose of TRC105 with PK samples collected at baseline and at least 1 time point on study
Measure: Mean (Full Range); unit: ug/mL
Groups:
- 10 mg/kg TRC105 + Pazopanib: All patients who received hybrid dose of 10 mg/kg TRC105 weekly followed by 15 mg/kg every other week in combination with 800 mg pazopanib daily
Arm/Group | 10 mg/kg TRC105 + Pazopanib
Number analyzed (Participants) | 6
ug/mL
  Cycle 2 Day 1 (4 weeks) trough PK concentrations | 124 [80 to 174]
  Cycle 2 Day 15 (6 weeks) trough PK concentrations | 86 [62 to 144]
  Cycle 3 Day 1 (8 weeks) trough PK concentrations: number analyzed (Participants) | 5
  Cycle 3 Day 1 (8 weeks) trough PK concentrations | 91 [73 to 121]
  Cycle 3 Day 15 (10 weeks) trough PK concentrations: number analyzed (Participants) | 4
  Cycle 3 Day 15 (10 weeks) trough PK concentrations | 80 [63 to 100]

5. Secondary Outcome: Number of Patients With and Without Development of Immunogenicity Antibodies (Phase 1 and 2)
Description: Anti-product antibody concentrations will be measured using validated ELISA methods. Anti-product antibody concentrations will be evaluated in the context of pharmacokinetic parameters and AE profiles.
Time Frame: 32 months
Population: All patients who received at least a portion of a dose of TRC105 with immunogenicity samples collected at baseline and at least 1 time point on study
Measure: Count of Participants; unit: Participants
Groups:
- 8 mg/kg TRC105 + Pazopanib: All patients who received TRC105 + Pazopanib TRC105: IV 8 mg/kg and Pazopanib: oral (800 mg)
- 10 mg/kg TRC105 + Pazopanib: All patients who received TRC105 + Pazopanib TRC105: IV 10 mg/kg and Pazopanib: oral (800 mg)
Arm/Group | 8 mg/kg TRC105 + Pazopanib | 10 mg/kg TRC105 + Pazopanib
Number analyzed (Participants) | 3 | 79
Participants
  Pt with treatment emergent ADA | 1 | 12
  Pt without treatment emergent ADA | 2 | 67

6. Secondary Outcome: Number of Patients With and Without Expression of Endoglin on Sarcoma Tissue (Phase 1 and 2)
Description: Expression will be determined by immunohistochemistry for each patient who received at least one dose of TRC105
Time Frame: 12 months
Population: All patients who received TRC105. Endoglin expression levels determined through archival tumor samples, which were drawn before dosing. Therefore dose levels combined.
Measure: Count of Participants; unit: Participants
Groups:
- TRC105 Plus Pazopanib: All patients in Phase 1b and Phase 2 portion of study who received TRC105 + Pazopanib TRC105: IV (8 mg/kg or 10 mg/kg). Pazopanib: oral (800 mg)
Arm/Group | TRC105 Plus Pazopanib
Number analyzed (Participants) | 66
Participants
  Tumor endoglin expression positive | 15
  Tumor endoglin expression negative | 51

7. Secondary Outcome: Objective Response Rate in Patients With Advanced Soft Tissue Sarcoma by RECIST 1.1
Description: The best response (CR, PR, SD or PD according to RECIST 1.1) for each patient (phase 1 and phase 2) with measurable disease who received at least one dose of TRC105 study drug
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 8 mg/kg TRC105 + Pazopanib | 10 mg/kg TRC105 + Pazopanib
Number analyzed (Participants) | 3 | 78
Participants
  Complete Response (CR) | 0 | 3
  Partial Response (PR) | 0 | 1
  Stable Disease (SD) | 3 | 43
  Progressive Disease (PD) | 0 | 27
  Not Evaluable | 0 | 4

8. Secondary Outcome: Progression Free Survival in a Cohort of Patients With Angiosarcoma (Phase 2)
Description: Time from screening to either first disease progression or death from any cause per RECIST version 1.1
Time Frame: 26 months
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | 10 mg/kg TRC105 + Pazopanib With Angiosarcoma
Number analyzed (Participants) | 9
months | 5.59 [2.1 to 15.78]

ADVERSE EVENTS:
Time Frame: Adverse events are collected for each patient from the time of informed consent through 28 days following the last dose of study drug. Patients were eligible for participation in the trial until they progressed. The longest duration of AE collection for a given patient was 34 months.
Arm/Group | 8 mg/kg TRC105 + Pazopanib | 10 mg/kg TRC105 + Pazopanib
All-Cause Mortality (participants affected / at risk) | 0/3 | 9/106
Serious Adverse Events (participants affected / at risk) | 0/3 | 9/106
Other Adverse Events (participants affected / at risk) | 3/3 | 106/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 8 mg/kg TRC105 + Pazopanib (N=3) | 10 mg/kg TRC105 + Pazopanib (N=106)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary Venous Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 8 mg/kg TRC105 + Pazopanib (N=3) | 10 mg/kg TRC105 + Pazopanib (N=106)
Fatigue (General disorders) | 2 | 80
Headache (Nervous system disorders) | 2 | 75
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 73
Nausea (Gastrointestinal disorders) | 2 | 66
Diarrhea (Gastrointestinal disorders) | 3 | 64
Vomiting (Gastrointestinal disorders) | 1 | 52
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 47
Hypertension (Vascular disorders) | 2 | 46
Anemia (Blood and lymphatic system disorders) | 1 | 45
Gingival Bleeding (Gastrointestinal disorders) | 2 | 40
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 37
Dysgeusia (Nervous system disorders) | 2 | 31
Pyrexia (General disorders) | 1 | 31
Stomatitis (Gastrointestinal disorders) | 1 | 25
Edema Peripheral (General disorders) | 0 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 22
Insomnia (Psychiatric disorders) | 1 | 22
Back Pain (Injury, poisoning and procedural complications) | 0 | 23
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 23
Flushing (Vascular disorders) | 0 | 22
Constipation (Gastrointestinal disorders) | 0 | 22
Weight Decreased (Investigations) | 0 | 21
Urinary Tract Infection (Infections and infestations) | 0 | 21
Palmar-Plantar Erythrodysaesthesia Syndrome (Infections and infestations) | 0 | 20
Dizziness (Nervous system disorders) | 1 | 19
Abdominal Pain (Gastrointestinal disorders) | 0 | 19
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 18
Rash (Skin and subcutaneous tissue disorders) | 0 | 17
Anxiety (Psychiatric disorders) | 0 | 17
Oral Pain (Gastrointestinal disorders) | 1 | 16
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 14
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 14
Hair Color Changes (Skin and subcutaneous tissue disorders) | 0 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 15
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 | 14
Asthenia (General disorders) | 0 | 15
Hypotension (Vascular disorders) | 0 | 14
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 14
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 13
Chills (General disorders) | 0 | 14
Gingival Pain (Gastrointestinal disorders) | 1 | 13
Erythema (Skin and subcutaneous tissue disorders) | 0 | 13
Migraine (Nervous system disorders) | 0 | 13
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 13
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 10
Hypokalemia (Metabolism and nutrition disorders) | 0 | 11
Aspartate Aminotransferase (Investigations) | 0 | 11
Influenza-like Illness (General disorders) | 0 | 11
Glossodynia (General disorders) | 0 | 11
Dry Mouth (Gastrointestinal disorders) | 1 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 10
Alanine Aminotransferase (Investigations) | 0 | 10
Oral Mucosal Exfoliation (Gastrointestinal disorders) | 1 | 9
Hypothyroidism (Endocrine disorders) | 0 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 10
Acute Kidney Injury (Renal and urinary disorders) | 0 | 9
Hyponatremia (Metabolism and nutrition disorders) | 0 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 8
Blood Bilirubin Increased (Investigations) | 1 | 8
Mouth Hemorrhage (Gastrointestinal disorders) | 0 | 9
Flatulence (Gastrointestinal disorders) | 0 | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 8
Depression (Psychiatric disorders) | 0 | 8
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 7
Mucosal Inflammation (General disorders) | 0 | 8
Malaise (General disorders) | 0 | 8
Chest Pain (General disorders) | 1 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Neuropathy Peripheral (Nervous system disorders) | 0 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 7
Lipase Increased (Investigations) | 0 | 7
Toothache (Gastrointestinal disorders) | 0 | 7
Gastroesophageal Reflux (Gastrointestinal disorders) | 0 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 6
Abdominal Upper Pain (Gastrointestinal disorders) | 0 | 7
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 6
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 4
Upper Respiratory Infection (Infections and infestations) | 2 | 4
Bronchitis (Infections and infestations) | 0 | 6
Disease Progression (General disorders) | 0 | 6
Oral Dysaesthesia (Gastrointestinal disorders) | 0 | 6
Vitreous Floaters (Eye disorders) | 0 | 6
Bradycardia (Cardiac disorders) | 0 | 6
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sinusitis (Infections and infestations) | 1 | 4
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Urinary Hesitation (Renal and urinary disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 3
Blood Calcium Decreased (Investigations) | 1 | 3
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 1
Loose Tooth (Gastrointestinal disorders) | 1 | 1
Visual Impairment (Eye disorders) | 1 | 3
Palpitations (Cardiac disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT01975519/Prot_SAP_000.pdf